CLINICAL TRIAL: NCT03418077
Title: Post-Exercise Cardiovascular Responses Following Energy Drink Consumption in Young, Healthy Adults
Brief Title: Post-Exercise Cardiovascular Responses Following Energy Drink Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: FDG20180006H
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: QTc Interval
MeSH Terms: interventions — Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- energy drink (Experimental): Participants will serve as their own controls and have repeated measures obtained to determine if there is a difference between the placebo-control and energy drink arms
  Interventions: Dietary Supplement: Energy Drink
- Placebo-control (Placebo Comparator): Participants will serve as their own controls and have repeated measures obtained to determine if there is a difference between the placebo-control and energy drink arms
  Interventions: Dietary Supplement: Placebo-control

INTERVENTIONS:
Dietary Supplement: Energy Drink — Participants will consume a randomly assigned single 24 oz can of an original flavor energy drink within a 30-minute period. Baseline ECG, HR, BP, blood sample and body weight will be obtained. Then perform a continuous, progressive treadmill or bicycle ergometry test until volitional exhaustion. ECG will be monitored continuously during exercise, rating of perceived exertion (RPE) will be recorded every minute of each workload increase. After completion of exercise, subject will remain standing on treadmill (or seated on ergometer) for 10 minutes while ECG, BP, HR and blood samples are obtained. Subsequent ECG measures will be obtained at 1,4,7 and 10 minutes. After 10 minutes, the subjects will be free to sit, stand or move quietly in the lab. During the 2-hour post exercise monitoring period, subject's ECG, HR, BP will be recorded at 30-minute intervals. Blood samples will be collected immediate upon cessation of exercise, at 1 and 2 hours post exercise
  Arms: energy drink
Dietary Supplement: Placebo-control — Participants will consume a randomly assigned single 24 oz can of control drink within a 30-minute period. Baseline ECG, HR, BP, blood sample and body weight will be obtained. Then perform a continuous, progressive treadmill or bicycle ergometry test until volitional exhaustion. ECG will be monitored continuously during exercise, rating of perceived exertion (RPE) will be recorded every minute of each workload increase. After completion of exercise, subject will remain standing on treadmill (or seated on ergometer) for 10 minutes while ECG, BP, HR and blood samples are obtained. Subsequent ECG measures will be obtained at 1,4,7 and 10 minutes. After 10 minutes, the subjects will be free to sit, stand or move quietly in the lab. During the 2-hour post exercise monitoring period, subject's ECG, HR, BP will be recorded at 30-minute intervals. Blood samples will be collected immediate upon cessation of exercise, at 1 and 2 hours post exercise
  Arms: Placebo-control

SUMMARY:
The purpose of this study is to determine the effects of consuming an original flavor energy drink on electrocardiographic (ECG) and hemodynamic responses during and after exercise in healthy subjects. The effect of drinking an energy drink on exercise performance will also be evaluated.

DETAILED DESCRIPTION:
The study will employ a double-blinded, randomized, crossover design to evaluate the cardiovascular (CV) effects of an energy drink during post-exercise recovery. Subjects who express interest in the study will be screen for eligibility. Those who are eligible will be consented. An inquire into usual caffeine intake to assess caffeine naïve or caffeine tolerant. Participants height, weight and race will be recorded. A resting 12-lead baseline ECG and blood pressure (BP) will be obtained to rule out CV anomalies. A cardiologist will review every baseline ECG and BP reading to rule out everything but a normal sinus rhythm and BP < 130/80 mmHg. Subjects who meet inclusion criteria and are approved by the cardiologist will be enrolled and allocated a randomized participant identification (ID) number. They will be given the "Participant Instruction Sheet"

Participants will be randomly assigned, blinded to consume a single 24 oz container of an energy drink or a 24 oz container of a control drink. Participants will serve as their own controls, so they will undergo testing in the experimental and control drink conditions, separated by 4 to 14 day. Each 24 oz control drink will be comprised of 585 ml of carbonated water, 30 ml of reconstituted lime juice and 105 ml of cherry flavoring. This control drink formula is identical to that used by Fletcher et al. (2017). The carbohydrate content of the 24 oz control drink is 81 g, which is the same as the 81 g per 24 oz energy drink. Participants will fast 12 hours, asked to refrain from vigorous exercised 24-hours, and abstain from caffeine consumption 48-hours prior to consuming a randomly assigned single 24 oz can of an original flavor energy drink within a 30-minute period. Investigator and participant will be blinded.

Subjects will be asked to visit either Heart, Lung and Vascular clinic or exercised physiology laboratory (CSUS subjects) twice, separated by 4-14 days to undergo testing. ECG electrodes will be placed on the upper torso and remain in place throughout the experiment. Baseline ECG, HR, BP, blood sample and body weight will be obtained. Catheter placement and blood draws will be performed by a registered clinical cardiopulmonary technician, registered nurse or a resident physician. Approximately 20 mil of blood will be taken at each time point.

Subjects will perform a continuous, progressive treadmill or bicycle ergometry test until volitional exhaustion. The treadmill test will begin with walking at 3.4 mph at 0% grade, then speed increased to 7 mph (males) or 6 mph (females) and grade increased by 2.5% every 2 minutes until > 85% ag-predicted maximum heart rate and volitional exhaustion has been reached. Subjects performing the ergometry test will being cycling at a resistance of 100 W for 2 minutes with the resistance increased by 25 W (males) or 15 W (females), each minute thereafter. Maximum HR will be calculated using the Tanaka formula (Tanaka et al., 2001). A 12-lead ECG will remain in place on subject and monitored continuously during exercise, and rating of perceived exertion (RPE) will be recorded every minute of each workload increase. After completion of exercise, subject will remain standing on treadmill (or seated on ergometer) for 10 minutes while ECG, BP, HR and blood samples are obtained. Subsequent ECG measures will be obtained at 1,4,7 and 10 minutes. After 10 minutes, the subjects will be free to sit, stand or move quietly in the lab. During the 2-hour post exercise monitoring period, subject's ECG, HR, BP will be recorded at 30-minute intervals. Blood samples for caffeine, taurine, L-carnitine, plasma free fatty acids, glucose and lactate will be collected immediate upon cessation of exercise, at 1 and 2 hours post exercise.

ELIGIBILITY:
Inclusion Criteria:

* Participants at David Grant Medical Center (DGMC): Healthy male and female, active duty military service members or Department of Defense (DoD) beneficiaries, who are eligible to receive care at DGMC. Participants at CSUS: Healthy male and female CSUS students.
* Ages 18-40 years old
* Participants must be willing to refrain from caffeine and energy drink use 48 hours prior to study days.

Exclusion Criteria:

* Cardiovascular risk factors: Heart rhythm other than normal sinus, history of atrial or ventricular arrhythmia, family history of premature sudden cardiac death before the age of 60, left ventricular hypertrophy, atherosclerosis, hypertension, palpitations, T-wave abnormalities, baseline corrected QT (QTc) interval greater than 440 milliseconds(msec). This will be determined on the ECG obtained during initial screening appointment, and reviewed by cardiologist and through the questionnaire responses of the participant.
* Blood pressure at initial screening appointment or at baseline on study Day 1 greater than 130/80
* Presence of any known medical condition, confirmed through participant interview. Examples of these are:

  * Hypertension
  * Thyroid disease
  * Type 1 or 2 diabetes mellitus
  * Recurrent headaches
  * Depression, currently receiving treatment (due to possible drug interactions)
  * Any psychiatric condition or neurological disorder
  * History of alcohol or drug abuse in the previous five years
  * Ever been diagnosed or told they have or had renal or hepatic dysfunction
* Concurrent use of any medication taken on a daily basis, to include herbal products or supplements. Daily basis is defined as greater than two days per week.
* Pregnant or lactating females will be excluded from participation with urine dipstick tests used to confirm pregnancy (pregnancy test performed before each treatment session).
* All non-English speaking / writing subjects and those that do not understand the study or consent process will be excluded from the study due to unavailability of medical qualified translator at all times during the study.
* If the subject refuses to sign the informed consent document or HIPAA Authorization, they will be excluded as well.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-07 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Change in QTc interval | 3 hours
  QTc interval will be obtained by 12-lead ECG at baseline (prior to consumption of study drink), after consuming the drink and immediately following exercise and at 1, 4, 7 and 10 min following exercise while standing, and again at 30-minute intervals for a total of 2 hours (after being seated for 5 minutes prior) after exercise. Measures will be obtained at two visits (i.e., one visit for the placebo drink and one visit for the energy drink), separated by 4 - 14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in systolic BP (SBP) | 3 hours
  SBP will be obtained at baseline (prior to consumption of study drink), after consuming the drink and immediately following exercise, and at again at 30-minute intervals for a total of 2 hours (after being seated for 5 minutes prior) after exercise. Measures will be obtained at two visits (i.e., one visit for the placebo drink and one visit for the energy drink), separated by 4 - 14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in diastolic BP (DBP) | 3 hours
  DBP will be obtained at baseline (prior to consumption of study drink), after consuming the drink and immediately following exercise, and again at 30-minute intervals for a total of 2 hours (after being seated for 5 minutes prior) after exercise. Measures will be obtained at two visits (i.e., one visit for the placebo drink and one visit for the energy drink), separated by 4 - 14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in heart rate (HR) | 3 hours
  HR will be obtained at baseline (prior to consumption of study drink), after consuming the drink and immediately following exercise, and at 1, 4, 7 and 10 minutes (while standing), and again at 30-minute intervals for a total of 2 hours after exercise (seated for 5 minutes prior). Measures will be obtained at two visits (i.e., one visit for the placebo drink and one visit for the energy drink), separated by 4 - 14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in blood parameters - caffeine | 3 hours
  Blood samples for caffeine will be obtained from a Teflon intravenous catheter that will remain in place throughout the duration of the experiment. Blood samples will be taken at baseline (prior to consumption of study drink); after consuming drink and immediately upon cessation of exercise, and at one-and two-hours following exercise. Blood samples will be obtained at two visits, (i.e., one visit for the energy drink and one visit for the placebo drink), separated by 4-14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and respective p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in blood parameters - taurine | 3 hours
  Blood samples for taurine will be obtained from a Teflon intravenous catheter that will remain in place throughout the duration of the experiment. Blood samples will be taken at baseline (prior to consumption of study drink); after consuming drink and immediately upon cessation of exercise, and at one-and two-hours following exercise. Blood samples will be obtained at two visits, (i.e., one visit for the energy drink and one visit for the placebo drink), separated by 4-14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and respective p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in blood parameters - L-caritine | 3 hours
  Blood samples for L-carnitine will be obtained from a Teflon intravenous catheter that will remain in place throughout the duration of the experiment. Blood samples will be taken at baseline (prior to consumption of study drink); after consuming drink and immediately upon cessation of exercise, and at one-and two-hours following exercise. Blood samples will be obtained at two visits, (i.e., one visit for the energy drink and one visit for the placebo drink), separated by 4-14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and respective p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in blood parameters - plasma free fatty acids | 3 hours
  Blood samples for plasma free fatty acids will be obtained from a Teflon intravenous catheter that will remain in place throughout the duration of the experiment. Blood samples will be taken at baseline (prior to consumption of study drink); after consuming drink and immediately upon cessation of exercise, and at one-and two-hours following exercise. Blood samples will be obtained at two visits, (i.e., one visit for the energy drink and one visit for the placebo drink), separated by 4-14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and respective p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in blood parameters - glucose | 3 hours
  Blood samples for glucose will be obtained from a Teflon intravenous catheter that will remain in place throughout the duration of the experiment. Blood samples will be taken at baseline (prior to consumption of study drink); after consuming drink and immediately upon cessation of exercise, and at one-and two-hours following exercise. Blood samples will be obtained at two visits, (i.e., one visit for the energy drink and one visit for the placebo drink), separated by 4-14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and respective p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in blood parameters - lactate | 3 hours
  Blood samples for lactate will be obtained from a Teflon intravenous catheter that will remain in place throughout the duration of the experiment. Blood samples will be taken at baseline (prior to consumption of study drink); after consuming drink and immediately upon cessation of exercise, and at one-and two-hours following exercise. Blood samples will be obtained at two visits, (i.e., one visit for the energy drink and one visit for the placebo drink), separated by 4-14 days. The values for each participant at each time point will be combined to obtain the means and standard deviations. The appropriate test statistic and respective p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data
Change in maximal exercise time to exhaustion | 3 hours
  After drink consumption, participants will perform a continuous, progressive treadmill or bicycle ergometer test until volitional exhaustion. Participants will be encouraged to perform their best during testing. Measures will be obtained on two days (i.e., one visit for the energy drink and one visit for the placebo drink), separated by 4 to 14 days. The values for each participant's maximal exercise time to exhaustion will be combined to obtain the means and standard deviations. The appropriate test statistic and p value will be reported to determine whether there was a statistically significant difference between the energy drink and placebo drink data

CONTACTS AND LOCATIONS:
Overall Officials: Troy D Chinevere, Principal Investigator — David Grant Medical Center
Locations (1):
- USAF David Grant Medical Center, Travis Air Force Base, California, United States